CLINICAL TRIAL: NCT03956290
Title: Time Restricted EATing (TREAT) Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Blandine Laferrere, Professor of Medicine, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAS3053
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Overweight and Obesity; Pre Diabetes
Keywords: Time restricted eating; Overweight; Obesity; Metabolic syndrome; Diabetes treated with metformin and/or diet and HbA1C< 7%; Pre Diabetes; Circadian rhythm
MeSH Terms: conditions — Overweight; Obesity; Glucose Intolerance; Intermittent Fasting; Metabolic Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TREAT pilot study (Experimental): Metabolically unhealthy overweight or obese potential participants who pass an in-person screen will enroll in a 2-week run-in period when they will use the app, to assess meal patterns under habitual living conditions.
  Interventions: Behavioral: TREAT pilot intervention

INTERVENTIONS:
Behavioral: TREAT pilot intervention — Participants will be asked to use the app and take pictures of everything they eat and drink, from the time they get up to the time they go to bed, regardless of size of meal/snacks/drink, for 2 weeks. This will generate data on their eating pattern and eating duration. Participants will be reminded through app, call or text by study staff based on personalized eating schedule. The sleep schedule will also be recorded.
  Other Names: TREAT

SUMMARY:
The TREAT Pilot is a 3 months open-label pilot study to examine the effect of restricting the duration of eating (Time Restricted EATing) in metabolically unhealthy adults with overweight or obesity. This pilot study will allow the investigator to collect preliminary data for the design of a larger study.

DETAILED DESCRIPTION:
Disruption of the circadian rhythm, caused by aging, obesity, shift work, or prolonged daily eating duration into hours normally reserved for sleep, is a recognized risk factor for impaired metabolism and cardiovascular disease risk. Mice with disrupted clock gene have dysmetabolism. Restricting the eating window in these mice improves their metabolism.

Data will be collected to examine the feasibility and effect of a lifestyle intervention, aiming to reduce body weight in metabolically unhealthy individuals with overweight and obesity. The TREAT pilot study employs the use of mobile application to document eating behavior, when, what and how much people eat. In addition, the participants will receive reminders and complete in-person study visits to monitor their eating and sleeping schedule.

ELIGIBILITY:
Inclusion Criteria:

* age: 45-73y old
* overweight or obesity with BMI ≥25.0 and ≤35.0 kg/m2
* pre-diabetes or diabetes only diet controlled (HbA1c <7%)
* elevated Blood Pressure (BP) 120-129/<80 mmHg or stage 1 high BP 130-139/80-89 mmHg, with clinical Atherosclerotic Cardiovascular Disease (ASCVD) or estimated 10-y Cardiovascular Disease (CVD) risk <10%
* having LDL cholesterol <150mg/dl
* no known sleep, psychiatric or food intake disorders
* in possession of a smart phone
* English-speaking
* must live in New York city geographical area and not have planned travel schedule interfering with the study

Exclusion Criteria:

* history or clinical evidence of condition that affect sleep
* significant organ system dysfunction/disease: diabetes, severe pulmonary, kidney or cardiovascular disease, and any evidence of active illness (e.g., fever)
* history of seizure disorder
* being on medications for diabetes, hypertension or dyslipidemia
* previous bariatric surgery
* history or current significant psychiatric disorder
* use dietary supplements and/or medications known to affect sleep, circadian rhythms or metabolic function
* smoking tobacco or using illegal or recreational drugs
* consume excessive alcohol (women: >14 drinks/wk; men: >21 drinks/wk)
* consume large amounts of caffeine daily (>2 cups of coffee or 8 oz caffeinated drinks per day)
* participate in intense exercise (causing heavy breathing and sweating, such as jogging) >2 d/wk for ≥35 min or moderate exercise (e.g., brisk walking) for >150 min/wk
* shift work
* extreme early and late chronotypes
* unwilling/unable to provide informed consent

Ages: 45 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
Percentage of participants logging | 3 months
  To measure the usage of app by recording the total number of days the participants logged in during study. Reported in percentage from 0 to 100% of time in use.
Percentage of patients who reduced eating duration by 4 hours | 3 months
  Change in eating duration from pre- to post-intervention will be calculated in from data collected in hours spent eating

SECONDARY OUTCOMES:
% weight loss achieved post-intervention | Baseline to 3 months
  Weight will be recorded and compared at baseline and 3 months.
Average time in duration of overnight fasting | 3 months
  Hours of overnight fasting will be recorded.
Average time in sleep duration | 3 months
  Hours of sleep each night will be recorded.
Adherence to using the app | 3 months
  Participants that completed daily food logs in app, and have days completed with correct eating duration.
% of participants who achieve ≥ 5% weight loss | Baseline to 3 months
  Weight will be recorded and compared at baseline and 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Blandine Laferrère, M.D., PhD., Principal Investigator — Columbia University
Locations (1):
- Obesity Nutrition Research Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Prasad M, Fine K, Gee A, Nair N, Popp CJ, Cheng B, Manoogian ENC, Panda S, Laferrere B. A Smartphone Intervention to Promote Time Restricted Eating Reduces Body Weight and Blood Pressure in Adults with Overweight and Obesity: A Pilot Study. Nutrients. 2021 Jun 23;13(7):2148. doi: 10.3390/nu13072148. PMID 34201442